CLINICAL TRIAL: NCT02672943
Title: The Role of Noradrenergic Network, and Its Association With Autonomous Dysfunction,Cerebral Autoregulation and microRNA in Parkinson Disease Before and After Medication and Rehabilitation Treatment
Brief Title: Parkinson Disease Before and After Medication and Rehabilitation Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRPG8D6031
Record Dates: First submitted 2015-04-01; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Autonomic nervous system; MicroRNA; Inflammation; Oxidative stress; noradrenergic network; Rehabilitation treatment
MeSH Terms: conditions — Parkinson Disease; Inflammation | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal (No Intervention): 30 normal volunteers with age, sex and BMI-match as control group
- treatment group (Active Comparator): The Rehabilitation treatment group will receive rehabilitation training once per day, 3 days per week, for 12 weeks. The duration of each session is about 1 hour. Participants will first receive relaxation exercises, positioning and self-stretch exercises (emphasizing on spinal mobility and flexor muscle groups of limbs and trunk) for 15 minutes. Then they will have balance training for 20 minutes. The investigators will use goal-directed tasks, such as different types of ball games, for balance training. At the end, participants will receive walking exercise for 20 minutes, and cool down exercises for 5 minutes.
  Interventions: Behavioral: Rehabilitation treatment
- non-treatment group (Sham Comparator): The group will not receive non-rehabilitation treatment, before and after the 12 weeks non-rehabilitation training, should accept MRI and Clinical assessments.
  Interventions: Other: non-rehabilitation treatment

INTERVENTIONS:
Behavioral: Rehabilitation treatment — The walking exercise will be aerobic with a Borg rating perceived exertion around 11-14 scales. Before and after the 12 weeks rehabilitation training, should accept MRI and Clinical assessments.
  Arms: treatment group
Other: non-rehabilitation treatment — The walking exercise will be aerobic with a Borg rating perceived exertion around 11-14 scales. Before and after the 12 weeks non-rehabilitation training, should accept MRI and Clinical assessments.
  Arms: non-treatment group

SUMMARY:
In this three-year project, our research teams are going to consecutively explore these important clinical, drug and physical rehabilitation treatment effects, noradrenergic network, autonomic dysfunction and microRNA signalling data as well as the correlations between them in early Parkinson Disease (PD) patients. The investigators hypothesize that the explorations of the above insights are unique and can provide an important source data for Taiwanese Parkinson Disease (PD).

DETAILED DESCRIPTION:
(1) 70 patients with PD. (2) 30 age and sex-match controls.

Methods:

-1st year To built up the biobank of 30 early PD patients (Hoehn and Yahr stage 1-3) and 30 health controls in all examination.

The PD patients will accept the MRI, autonomic dysfunction, and peripheral microRNA examination and their correlations among each other at least 12 hours after the least medication.

-2nd year Second year, the investigators will follow-up the 30 PD patients enrolled in the 1st years.

The PD patients will receive studies to evaluate the pharmacokinetics effect before medication, including MRI, autonomic dysfunction, and peripheral microRNA examination.

-3rd year the investigators will study the rehabilitation effect in PD (3 days per week, for 12 weeks).

30 PD with rehabilitation and 30 PD without rehabilitation will be enrolled and compared their difference in MRI study, autonomic dysfunction, and peripheral microRNA examination before and after 3 month follow-up.

Goals

1. To define the effect of norepinephrine network to autonomic dysfunction in PD
2. To define the effect of peripheral microRNA level to norepinephrine network in PD
3. To associate drug/physical rehabilitation effect to alteration of norepinephrine network, autonomic dysfunction, and peripheral microRNA and their interactions to striatal dopaminergic network in PD.
4. According to previous results, to verify the role of norepinephrine network and autonomic dysfunction in long-term PD evolution.

ELIGIBILITY:
Inclusion Criteria:

* In this study, the patients should be 40-75 years of age and identified as PD. PD patients with an early clinical stage (Hoehn and Yahr stage 1-3) will be enrolled in this study. The informed written consent which is approved by Ethics Committee of our hospital will be obtained from the patient or their family.

Exclusion Criteria:

* Patients with the following conditions are excluded:

  1. Atherosclerotic narrowing on intracranial and extracranial vessels (>50% stenosis) with or without evidence of old cerebral infarctions, coronary artery diseases status post percutaneous transluminal coronary angioplasty or bypass surgery and renal failure requiring hemodialysis or peritoneal dialysis
  2. Moderate to severe heart failure (NYHA class III and IV).
  3. Central or peripheral disorders known to affect autonomic nervous systems.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Neuroimage | 12 weeks
  Conventional MRI, Rest function MRI Image Data Preprocessing, Assessment of cerebral blood flow with Arterial Spin Labeling (ASL) MRI and Chemical Exchange Saturation Transfer

SECONDARY OUTCOMES:
Physical Rehabilitation_1 | 12 weeks
  Unified Parkinson's Disease Rating Scale
Physical Rehabilitation_2 | 12 weeks
  Walking speed by self-selected gait speed over 10 m
Physical Rehabilitation_3 | 12 weeks
  Walking endurance, by using the 6-minute walk test
Physical Rehabilitation_4 | 12 weeks
  Static and dynamic balance control, by using Biodex Balance System and Timed Up and Go test
Biochemical Analysis | 18 months
  interval change of serum MicroRNA level (increase of decrease)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsien Lu, M.D., Study Director — Chang Gung Memorial Hospital; Jen-Wen Hung, M.D., Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No